CLINICAL TRIAL: NCT06084442
Title: Evaluation of The Techniques of Lateral Rectus Muscle Combined Recession With Hang Back and Combined Recession With Z-Tenotomy in Correcting Large-Angle Exotropia
Brief Title: Evaluation of The Techniques in Correcting Large-Angle Exotropia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Basma Gamal Mohamed Ahmed Sayed Ahmed, Assistant lecturer, Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Large-Angle Exotropia
Record Dates: First submitted 2023-10-09; First posted 2023-10-16 (Actual); Last update posted 2023-10-16 (Actual); Status verified 2023-10

CONDITIONS: Exotropia; Evaluation of Surgical Techniques in Correcting Exotropia
MeSH Terms: conditions — Exotropia

STUDY DESIGN:
Intervention Model Description: Patients will be divided into 2 groups:
  * Group (A): Patients will undergo combined LR recession 7mm and hang back technique.
  * Group (B): Patients will undergo combined LR recession 7mm and Z-tenotomy technique.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- combined lateral rectus muscle recession 7mm and hang back technique. (Active Comparator): The technique of combined LR recession 7mm and hang back technique:
  A. The muscle is exposed in the usual manner and locking suture is passed through full thickness of the LR muscle using nonabsorbable ethibond suture.
  B. The muscle is cut from its insertion site. C. Marking the sclera for the rectus muscle recession. a Measurement from the limbus, or b measurement from the original insertion site.
  D. Passage of the needles in the sclera using the "crossed swords" Technique E. The muscle has been pulled up to its new insertion point and the sutures have been tied and cut and the remainder of the procedure is identical to the standard hang-back method.
  The
  Interventions: Procedure: Evaluation of The Techniques of Lateral Rectus Muscle Combined Recession with Hang Back and Combined Recession with Z-Tenotomy in Correcting Large-Angle Exotropia
- combined lateral rectus muscle recession 7mm and Z- tenotomy technique. (Active Comparator): The technique of lateral rectus muscle Z-tenotomy:
  A. The muscle is exposed in the usual manner and two hemostats are each placed 80% of the way across the muscle (or tendon) from opposite borders. The hemostats are placed 3 or 4 mm apart.
  B. The posterior hemostat is removed, and scissors are used to cut across the muscle in the crushed area. By cutting the muscle in the crushed area, bleeding is kept to a minimum.
  C. The hemostat nearer the insertion is removed, and the muscle is cut along the crushed area using small snips with scissors.
  D. lengthening of the muscle will occur. Any bleeding is controlled with pressure.
  E. After the distal myotomy has been performed, in a very tight muscle, a No. 15 Bard Parker blade can be used to divide the tendon fibers, cutting against the muscle hook. This can be accomplished with a scraping motion with the knife blade at nearly right angles to avoid scleral perforation.
  Interventions: Procedure: Evaluation of The Techniques of Lateral Rectus Muscle Combined Recession with Hang Back and Combined Recession with Z-Tenotomy in Correcting Large-Angle Exotropia

INTERVENTIONS:
Procedure: Evaluation of The Techniques of Lateral Rectus Muscle Combined Recession with Hang Back and Combined Recession with Z-Tenotomy in Correcting Large-Angle Exotropia — Patients will be divided into 2 groups:
  * Group (A): Patients will undergo combined LR recession 7mm and hang back technique.
  * Group (B): Patients will undergo combined LR recession 7mm and Z-tenotomy technique.

SUMMARY:
The aim of this study is to evaluate the techniques of combined lateral rectus muscle recession with hang back and combined lateral rectus muscle recession with z-tenotomy in correcting large-angle exotropia.

DETAILED DESCRIPTION:
Strabismus was defined as any heterotropia at near or distance fixation, or both, on cover testing. Micro strabismus was known as a deviation of fewer than 10 prism diopters (PD). Different studies have defined large angle deviation as 35 Δ , 40 Δ, 50 Δ and 60 Δ.

Studies revealed that during the first decade of life, exotropia is most prevalent with intermittent exotropia and convergence insufficiency are the most frequent. Exotropic deviations include exophoria, infantile exotropia, intermittent exotropia, sensory exotropia and consecutive exotropia.

Large-angle constant exotropia has a negative impact on the patients and surgical treatment of exodeviations improves the patient's psychosocial functioning. Hence, many surgical techniques have been described for management of exotropia, including bilateral lateral rectus recessions or recess/resect procedures. Botulinum toxin injection combined with recession-resection procedures was used as another surgical technique.

As a fact large-angle exotropia usually requires greater amounts of surgery, often a surgery on a greater number of extraocular muscles. Hence, 3 or 4 horizontal muscle surgery was performed for correcting large angle exotropia. Single-staged three horizontal muscles surgery for large angle intermittent exotropia has been more successful.

Recently, medial rectus muscle surgery as bilateral medial rectus resection for primary large-angle exotropia has been used with successful results. A successful outcome of surgery was defined as deviation within 10 prism diopters for both distance and near.

Moreover, hang-back loop suspension surgical technique can be performed for lateral rectus (LR) muscle recession. This technique can offer potential advantages over the conventional rectus muscle recession, including better exposure of the site of scleral sutures, lower risk of scleral perforation , shorter procedure duration and lower postoperative induced astigmatism.

On the other hand, the hang-back recession has some limitations as a potential unpredictability in surgical outcomes.Although previous reports suggest that the hang-back technique for LR recession for exotropia results in poorer surgical success and may require a different surgical dosage, another study proved that the hang-back surgical technique was as effective as conventional LR recession surgery for children with exotropia.

Furthermore, many studies were performed on Z-tenotomy technique as an alternative procedure for muscle weakening. This technique was applied for superior oblique muscle in cases with mild to moderate over depression in adduction with success rate 90%. An Other study has revealed that z-tenotomy up to 50% progressively reduces extraocular tendon force transmission, but Z-tenotomy of ≥50% is biomechanically equivalent in vitro to complete tenotomy.

In the past it was thought that muscle recessions with the muscle placed behind the anatomical equator of the globe would cause limitation of ocular rotation. Postoperative abduction limitation is one of the main problems in large recession and/or resection for primary and recurrent exotropia with large angle. It is generally thought that keeping the lateral rectus recession to no more than 8 mm prevents this complication. However, several studies revealed that large amounts of recession can be done without causing significant ocular movement limitation.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from large angle exotropia; defined, in this study, as an angle of deviation ≥ 40 prism diopters (PD).

Exclusion Criteria:

1. Patients suffering from exotropia with angle < 40 prism diopters (PD).
2. Patient with paralytic strabismus.
3. Patient with restrictive strabismus.
4. Patient with combined vertical and horizontal deviation.
5. Patients with previous strabismus surgery.
6. Patients who had previously been administered botulinum toxin A.
7. Patient refusal.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-10 (Estimated); Primary Completion 2024-03 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
sucessful alignment | Follow up period of 6 month from the time of initial surgery. All patients will be examined at one week, one month, 3 month and 6 months.
  Successful motor alignment will be defined as orthotropia or ≤ 10 Δ Exotropia or Esotropia at 6 m distance with spectacle correction worn at 6 months. Successful sensory alignment will be by achievement of fusion and moderate or good stereoacuity postoperatively.

CONTACTS AND LOCATIONS:
Overall Officials: El-Sayed Samir Arafa, MD, Study Director — Tanta University; Amr Mahmoud Awara, MD, Study Director — Tanta University; Heba Mohamed Shafik, MD, Study Director — Tanta University

REFERENCES:
- [Background] Livir-Rallatos G, Gunton KB, Calhoun JH. Surgical results in large-angle exotropia. J AAPOS. 2002 Apr;6(2):77-80. doi: 10.1067/mpa.2002.122059. PMID 11997802
- [Background] Chen JH, Morrison DG, Donahue SP. Three and Four Horizontal Muscle Surgery for Large Angle Exotropia. J Pediatr Ophthalmol Strabismus. 2015 Sep-Oct;52(5):305-10. doi: 10.3928/01913913-20150609-02. Epub 2015 Jun 15. PMID 26098544
- [Background] Chung AK, Rehman SU, Bradbury JA. Comparison of modified anchored "hang-back technique (HBT)" with conventional HBT in bimedial rectus recession. J AAPOS. 2005 Jun;9(3):234-9. doi: 10.1016/j.jaapos.2005.02.011. PMID 15956942
- [Background] Betts C, Olitsky S. Corneal astigmatic effects of conventional recession vs suspension recession ("hang-back") strabismus surgery: a pilot study. Binocul Vis Strabismus Q. 2006;21(4):211-3. PMID 17069557
- [Background] Orlin A, Mills M, Ying GS, Liu C. A comparison of hang-back with conventional recession surgery for exotropia. J AAPOS. 2007 Dec;11(6):597-600. doi: 10.1016/j.jaapos.2007.06.001. Epub 2007 Oct 24. PMID 17920319
- [Background] Shin A, Yoo L, Demer JL. Biomechanics of superior oblique Z-tenotomy. J AAPOS. 2013 Dec;17(6):612-7. doi: 10.1016/j.jaapos.2013.09.004. PMID 24321425